CLINICAL TRIAL: NCT02425241
Title: A Randomised Double-blind, Placebo-controlled Phase I/IIa Trial to Investigate the Effect of Depletion of Serum Amyloid P Component (SAP) on the Immune Response to DNA Vaccination in Healthy Male Volunteers
Brief Title: Depletion of Serum Amyloid P Component to Enhance the Immune Response to DNA Vaccination
Acronym: HIV-CORE003
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); University of Oxford (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HIV-CORE003; 2012-004052-11 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2015-04-23 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: Vaccine; DNA; HIV-1; Serum amyloid P component (SAP); Clinical trial; Vaccination; Prophylaxis; Adult male
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPHPC (Experimental): CPHPC infusion over 26 hours to deplete SAP at weeks 0,4 and 8. pSG2.HIVconsv DNA vaccine 4 mg at weeks 0, 4 and 8 after 24 hours of CPHPC infusion.
  ChAdV63.HIVconsv booster vaccine 5 x 10^10 vp at week 12. MVA.HIVconsv booster vaccine 2 x 10^8 pfu at week 20
  Interventions: Biological: pSG2.HIVconsv DNA vaccine; Biological: ChAdV63.HIVconsv booster vaccine; Biological: MVA.HIVconsv booster vaccine; Drug: CPHPC
- 0.9% w/v saline solution (Placebo Comparator): Placebo (normal saline) infusion over 26 hours at weeks 0,4 and 8. pSG2.HIVconsv DNA vaccine 4 mg at weeks 0, 4 and 8 after 24 hours of placebo infusion.
  ChAdV63.HIVconsv booster vaccine 5 x 10^10 vp at week 12. MVA.HIVconsv booster vaccine 2 x 10^8 pfu at week 20
  Interventions: Biological: pSG2.HIVconsv DNA vaccine; Biological: ChAdV63.HIVconsv booster vaccine; Biological: MVA.HIVconsv booster vaccine; Other: Placebo

INTERVENTIONS:
Biological: pSG2.HIVconsv DNA vaccine — pSG2.HIVconsv DNA 4 mg at weeks 0, 4 and 8.
Biological: ChAdV63.HIVconsv booster vaccine — ChAdV63.HIVconsv 5 x 10^10 vp at week 12.
Biological: MVA.HIVconsv booster vaccine — MVA.HIVconsv 2 x 10^8 pfu at week 20
Drug: CPHPC — 40 mg CPHPC IV infusion for 26 hours at weeks 0, 4 and 8 during which pSG2.HIVconsv is administered after 24 hours.
  Other Names: (R)-1-[6-[(R)-2-carboxy-pyrrolidin-1-yl]-6-oxohexanoyl] pyrrolidine-2-carboxylic acid
  Arms: CPHPC
Other: Placebo — Placebo IV infusion for 26 hours at weeks 0, 4 and 8 during which pSG2.HIVconsv is administered after 24 hours.
  Other Names: 0.9% saline
  Arms: 0.9% w/v saline solution

SUMMARY:
This is a clinical proof-of-concept (PoC) study of DNA vaccination after SAP depletion. The investigators will measure the immune responses to DNA vaccination against HIV-1 in healthy adult male volunteers, comparing a group in whom SAP has been completely depleted at the time of DNA vaccination and a control group vaccinated without SAP depletion.

DETAILED DESCRIPTION:
Vaccination is one of the most important achievements of medicine. Injection of modified germs, or materials from them, induces protective immunity against the infections which they cause. Successful immunisation induces a protective immune response against particular component(s) of the target germ, the so-called immunogen(s). For some diseases the immunogens are not known and for others they are difficult and expensive to produce, transport and administer, for example influenza vaccine must be produced in millions of chicken eggs. A very attractive potential solution is to inject the deoxyribose nucleic acid (DNA) gene encoding the immunogen rather than the immunogen itself. In this process, known as DNA vaccination, the DNA enters cells, predominantly at the site of injection, and causes them to produce the immunogen locally within the body. DNA vaccination works well and stimulates excellent protective immunity against a variety of different infections, and even some cancers, in mice, horses, dogs, rabbits and pigs. But in humans and other primates, and in cows and sheep, the immune response to DNA vaccination is very feeble. Despite enormous academic and pharmaceutical industry efforts, the reasons for this failure have not been understood or overcome. The investigators previously discovered that a protein in human blood, known as serum amyloid P component (SAP), is the only normal blood protein which binds strongly to DNA. The investigators have now found that, in each of the animal species in which DNA vaccination is effective, this protein is either absent or, if it is present, it binds only weakly to DNA. In contrast, nonhuman primates, cows and sheep share with humans the presence of SAP proteins which strongly bind to DNA. The investigators believe that binding of DNA by SAP may be responsible for blocking induction of immune responses by DNA and that removal of SAP may overcome this inhibition. SAP contributes to important human diseases, amyloidosis and Alzheimer's disease, and the investigators have previously developed a drug, (R)-1-[6-[(R)-2-carboxy-pyrrolidin-1-yl]-6-oxohexanoyl]pyrrolidine-2-carboxylic acid (CPHPC), which safely removes almost all SAP from the blood in humans. Another laboratory has recently reported that the presence of human SAP inhibits DNA vaccination in mice and that this effect is reversed by the investigators drug, CPHPC. These observations confirm the investigators hypothesis. The investigators now propose to undertake the first human clinical study of DNA vaccination after SAP depletion. The investigators will measure the immune responses to human immunodeficiency virus (HIV)-1 DNA vaccination in 40 healthy adult men, comparing a group in whom SAP has been completely depleted at the time of DNA vaccination and a control group vaccinated without SAP depletion. The investigators predict that SAP depletion at the time of DNA vaccination will enhance the immune response.

Development of an effective, accessible vaccine is the only realistic hope for halting the human immunodeficiency virus type 1 (HIV-1)/AIDS epidemic. Ideally, such a vaccine should induce broadly neutralizing antibodies and effective T cells at the same time. Both of these goals face substantial and very different challenges, with one major roadblock in common: the enormous HIV-1 genome plasticity, i.e. ability to change and escape immune responses. There is a need to develop vaccines which may be used both prophylactically and therapeutically to either prevent HIV-1 acquisition, control its replication without HAART and/or eventually eradicated the virus from the body completely.

The approach taken in this clinical study aims to overcome the antigenic variation of HIV-1 by focusing induced T cell responses on the functionally conserved regions of HIV-1 proteins, which HIV-1 cannot change without a significant cost to its fitness. Thus, the HIVconsv immunogen is a chimaeric protein assembled from the 14 most conserved regions of the HIV-1 proteome alternating among the four most common HIV-1 clades: A, B, C and D. The gene coding for HIVconsv was made synthetically and was inserted into three safe non-replicating vaccine vectors: plasmid DNA to construct pSG2.HIVconsv, attenuated chimpanzee adenovirus (ChAdV63) to construct ChAdV63.HIVconsv and recombinant modified vaccinia virus Ankara (MVA) to construct MVA.HIVconsv. These three vectors facilitate delivery of the immunogen gene into host cells, which then express the HIVconsv protein and initiate a series of processes leading to the presentation of HIVconsv-derived peptides to the cells of the host immune system and induction of the HIVconsv-specific host T cell responses.

Volunteers will receive the vaccine candidates ChAdV63.HIVconsv (C), MVA.HIVconsv (M) and pSG2.HIVconsv DNA (D) in a DDDCM regimen at weeks 0, 4, 8, 12 and 16. CPHPC or placebo is given by 26 hours infusion prior to the pSG2.HIVconsv vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, as assessed by a medical history, physical examination and laboratory tests.
* Aged at least 18 years on the day of screening and no greater than 50 years on the day of the first vaccination.
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
* In the opinion of the Chief Investigator (CI) or designee, the volunteer has understood the information provided and is able to provide written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Willing to undergo HIV-1 testing, HIV-1 counselling and receive HIV-1 test results.
* If heterosexually active male; willing to use an effective method of contraception from the day of the first vaccination until six weeks after the last vaccination.
* Willing to forgo donating blood during the study.

Exclusion Criteria:

* None.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
vaccine safety (Proportion of volunteers who develop a grade 3 or grade 4 local reaction/ grade 3 or 4 systemic reaction) | 20 weeks
  Proportion of volunteers who develop a grade 3 or grade 4 local reaction. Proportion of volunteers who develop a grade 3 or grade 4 systemic reaction.
vaccine immunogenicity (T cell responses will be determined initially by interferon-gamma enzyme-linked immunospot assay) | 20 weeks
  T cell responses will be determined initially by interferon-gamma enzyme-linked immunospot assay.

CONTACTS AND LOCATIONS:
Overall Officials: Julian D Gillmore, MBBS, Principal Investigator — University College, London
Locations (1):
- National Amyloidosis Centre, London, England, United Kingdom

REFERENCES:
- [Derived] Borthwick NJ, Lane T, Moyo N, Crook A, Shim JM, Baines I, Wee EG, Hawkins PN, Gillmore JD, Hanke T, Pepys MB. Randomized phase I trial HIV-CORE 003: Depletion of serum amyloid P component and immunogenicity of DNA vaccination against HIV-1. PLoS One. 2018 May 17;13(5):e0197299. doi: 10.1371/journal.pone.0197299. eCollection 2018. PMID 29772028